CLINICAL TRIAL: NCT05177848
Title: Comparison of the Substitution Between Different Tobacco/Nicotine Products as a Function of Tobacco-user Type
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Medical University of South Carolina (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roberta Freitas-Lemos, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB #21-1046; 5P01CA200512 (NIH)
Record Dates: First submitted 2021-12-14; First posted 2022-01-05 (Actual); Results first posted 2024-09-26 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-08

CONDITIONS: Cigarette Smoking; Nicotine Vaping
MeSH Terms: conditions — Cigarette Smoking; Vaping

STUDY DESIGN:
Intervention Model Description: Participants will complete seven Experimental Tobacco Marketplace conditions. Conventional cigarette price will be parametrically increased, and the purchasing of alternative products measured. Alternative products (i.e. nicotine vaping products, heated tobacco products and nicotine pouches) will be available at different prices in separate conditions (i.e., ½ market price, market price, and 2x market price).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exclusive cigarette smokers (Experimental): Exclusive cigarette smokers will be recruited and will be exposed to all of the conditions described in the intervention section.
  Interventions: Other: All nicotine/ tobacco products at market price; Other: Nicotine vaping products at 1/2 market price; Other: Nicotine vaping products at 2x market price; Other: Heated tobacco products at 1/2 market price.; Other: Heated tobacco products at 2x market price.; Other: Nicotine pouch products at 1/2 market price.; Other: Nicotine pouch products at 2x market price.
- Dual cigarette/ nicotine vaping product users (Experimental): Dual cigarette and nicotine vaping product users will be recruited and will be exposed to all of the conditions described in the intervention section.
  Interventions: Other: All nicotine/ tobacco products at market price; Other: Nicotine vaping products at 1/2 market price; Other: Nicotine vaping products at 2x market price; Other: Heated tobacco products at 1/2 market price.; Other: Heated tobacco products at 2x market price.; Other: Nicotine pouch products at 1/2 market price.; Other: Nicotine pouch products at 2x market price.

INTERVENTIONS:
Other: All nicotine/ tobacco products at market price — Nicotine/tobacco products available in the Experimental Tobacco Marketplace at market price. Note that all participants will complete all the specified conditions.
Other: Nicotine vaping products at 1/2 market price — Availability of nicotine vaping products in the Experimental Tobacco Marketplace at 1/2 market price. Other nicotine/tobacco products at market price. Note that all participants will complete all the specified conditions.
Other: Nicotine vaping products at 2x market price — Availability of nicotine vaping products in the Experimental Tobacco Marketplace at 2x market price. Other nicotine/tobacco products at market price. Note that all participants will complete all the specified conditions.
Other: Heated tobacco products at 1/2 market price. — Availability of heated tobacco products in the Experimental Tobacco Marketplace at 1/2 market price. Other nicotine/tobacco products at market price. Note that all participants will complete all the specified conditions.
Other: Heated tobacco products at 2x market price. — Availability of heated tobacco products in the Experimental Tobacco Marketplace at 2x market price. Other nicotine/tobacco products at market price. Note that all participants will complete all the specified conditions.
Other: Nicotine pouch products at 1/2 market price. — Availability of heated tobacco products in the Experimental Tobacco Marketplace at 1/2 market price. Other nicotine/tobacco products at market price. Note that all participants will complete all the specified conditions.
Other: Nicotine pouch products at 2x market price. — Availability of heated tobacco products in the Experimental Tobacco Marketplace at 2x market price. Other nicotine/tobacco products at market price. Note that all participants will complete all the specified conditions.

SUMMARY:
This study will investigate the relative appeal (abuse liability) of novel tobacco products, how the appeal is modulated by relative price, user type, and how novel products may substitute for one another.

DETAILED DESCRIPTION:
An important aim of tobacco control is to reduce demand for the most harmful products. Therefore, a priori knowledge of substitutability across novel and widely used tobacco products may forecast the impact of policies on product switching. This study will use a novel method, the Experimental Tobacco Marketplace (ETM), to characterize the relative substitutability and appeal (abuse liability) of tobacco products (e.g., conventional cigarettes, nicotine vaping products [NVP], heated tobacco products [HTP], and nicotine pouch products [NPP]), and how the appeal is modulated by relative price and user type. Exclusive cigarette smokers and dual cigarette/NVP users, stratified by age, will complete multiple scenarios in the ETM.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent
* Be at least 21 years of age or older
* Provide a breath sample for measuring carbon monoxide (CO ≥ 8 ppm)
* Stable tobacco use patterns for at least three months
* Be willing to sample NVPs, HTPs, and NPPs
* For exclusive cigarette smokers: smoke at least 10 cigarettes daily and do not use NVPs regularly (no more than 9 times in the last month)
* For dual cigarette/NVP users: smoke at least 5 cigarettes daily and use NVPs for at least 3 times in a week (report use of closed nicotine salt system)

Exclusion Criteria:

* Have plans to move out of the area
* Have a serious or unstable physical or mental health condition
* Taking a tobacco cessation medication or medication that interferes with nicotine metabolism, motivation or reinforcement
* Report concrete, immediate plans to alter/quit using their usual nicotine products at the beginning of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren K Bickel, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
The study team will share de-identified data upon request.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants are assigned to exclusive smokers or dual cigarette/nicotine vaping product users groups based on the screening form.
Groups:
- Exclusive Cigarette Smokers: Exclusive smokers will be recruited and exposed to all conditions described in the intervention section.
  All nicotine/ tobacco products at market price: Nicotine/tobacco products available in the Experimental Tobacco Marketplace (ETM) at market price.
  Nicotine vaping products at 1/2 market price: Availability of nicotine vaping products in the ETM at 1/2 market price. Other nicotine/tobacco products at market price.
  Nicotine vaping products at 2x market price: Availability of nicotine vaping products in the ETM at 2x market price. Other nicotine/tobacco products at market price.
  Heated tobacco products at 1/2 market price.: Availability of heated tobacco products in the ETM at 1/2 market price. Other nicotine/tobacco products at market price.
  Heated tobacco products at 2x market price.: Availability of heated tobacco products in the ETM at 2x market price. Other nicotine/tobacco products at market price.
  Nicotine pouch products at 1/2 market price.: Availability of heated tobacco products in the ETM at 1/2 market price. Other nicotine/tobacco products at market price.
  Nicotine pouch products at 2x market price.: Availability of heated tobacco products in the ETM at 2x market price. Other nicotine/tobacco products at market price.
- Dual Cigarette/ Nicotine Vaping Product Users: Dual cigarette and nicotine vaping product users will be recruited and exposed to all conditions described in the intervention section.
  All nicotine/ tobacco products at market price: Nicotine/tobacco products available in the Experimental Tobacco Marketplace (ETM) at market price. Note that all participants will complete all the specified conditions.
  Nicotine vaping products at 1/2 market price: Availability of nicotine vaping products in the ETM at 1/2 market price. Other nicotine/tobacco products at market price.
  Nicotine vaping products at 2x market price: Availability of nicotine vaping products in the ETM at 2x market price. Other nicotine/tobacco products at market price.
  Heated tobacco products at 1/2 market price.: Availability of heated tobacco products in the ETM at 1/2 market price. Other nicotine/tobacco products at market price.
  Heated tobacco products at 2x market price.: Availability of heated tobacco products in the ETM at 2x market price. Other nicotine/tobacco products at market price.
  Nicotine pouch products at 1/2 market price.: Availability of heated tobacco products in the ETM at 1/2 market price. Other nicotine/tobacco products at market price.
  Nicotine pouch products at 2x market price.: Availability of heated tobacco products in the ETM at 2x market price. Other nicotine/tobacco products at market price.
Period: Overall Study
Arm/Group | Exclusive Cigarette Smokers | Dual Cigarette/ Nicotine Vaping Product Users
Started | 29 | 31
Completed | 26 | 26
Not Completed | 3 | 5
Not completed — Lost to Follow-up | 1 | 4
Not completed — Discontinued | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exclusive Cigarette Smokers | Dual Cigarette/ Nicotine Vaping Product Users | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.19 (10.63) | 37.00 (9.98) | 36.10 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 15 | 10 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 24 | 25 | 49
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 22 | 21 | 43
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Number of cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes smoked per day] | 18.22 (7.31) | 19.74 (8.97) | 18.97 (8.14)

OUTCOME MEASURES:

1. Primary Outcome: Nicotine/Tobacco Products Substitution
Description: Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM) with cigarettes increasing in price. Other product prices in the ETM will depend on the experimental condition. The degree to which other nicotine/tobacco products substitute for conventional cigarettes as a function of novel product (e.g. nicotine vaping products, heated tobacco products, nicotine pouch products) prices will be assessed.
  To obtain estimates of substitution of price-constant products in the different ETM conditions, the investigators will use ordinary least squares regression to model the relationship of the price-manipulated product to predict total quantity purchased of the price-constant product.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mg of nicotine purchased
Arm/Group | Exclusive Cigarette Smokers | Dual Cigarette/ Nicotine Vaping Product Users
Number analyzed (Participants) | 26 | 26
mg of nicotine purchased
  Control | 12.11 (51.66) | 4.82 (25.93)
  HTP 1/2 | 25.28 (45.78) | 17.08 (22.07)
  HTP 2 | 19.70 (43.92) | 10.73 (24.88)
  NPP 1/2 | 20.77 (52.88) | 11.06 (28.00)
  NPP 2 | 16.36 (50.81) | -1.09 (27.51)
  NVP 1/2 | 11.62 (118.50) | -0.68 (81.91)
  NVP 2 | 24.56 (39.38) | 11.58 (26.46)
Statistical Analysis 1: Comparison: Exclusive Cigarette Smokers vs Dual Cigarette/ Nicotine Vaping Product Users; Test type: Other; p = 0.9793, Mixed Models Analysis — A linear mixed effects model tested the interaction between group and condition on the rate of substitution Results: Condition: X2(6) = 4.30, p = 0.64 Group: X2(1) 0.22, p = 0.64 Condition:Group: X2(6) = 1.15, p = 0.98

2. Primary Outcome: Cigarette Demand
Description: Participants will complete purchasing trials in an Experimental Tobacco Marketplace (ETM) with cigarettes increasing in price. Other product prices in the ETM will depend on the experimental condition. The degree to which other nicotine/tobacco products substitute for conventional cigarettes as a function of novel product (e.g. nicotine vaping products, heated tobacco products, nicotine pouch products) prices will be assessed.
  To obtain dependent measures of demand, participants' purchasing of the price-manipulated commodity in the ETM task will be fit to a modified exponential equation to quantify the relationship between the price of each commodity and purchasing: Q=Q0*10k(exp(-αQ0C)-1) where Q is purchasing of the commodity, C is the price, Q0 is the derived initial purchasing without cost constraints (demand intensity), k is the span of the function in logarithmic units, and α is the demand elasticity.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mg of nicotine purchased
Arm/Group | Exclusive Cigarette Smokers | Dual Cigarette/ Nicotine Vaping Product Users
Number analyzed (Participants) | 26 | 26
mg of nicotine purchased
  Control | 212.39 (206.92) | 193.58 (258.37)
  HTP 1/2 | 221.66 (235.08) | 163.28 (170.31)
  HTP 2 | 186.03 (206.94) | 231.96 (391.03)
  NPP 1/2 | 229.45 (225.12) | 186.18 (200.50)
  NPP 2 | 225.77 (217.11) | 163.71 (225.14)
  NVP 1/2 | 187.58 (205.34) | 184.45 (229.39)
  NVP 2 | 198.93 (197.99) | 237.64 (309.73)
Statistical Analysis 1: Comparison: Exclusive Cigarette Smokers vs Dual Cigarette/ Nicotine Vaping Product Users; Test type: Other; p = 0.29, Mixed Models Analysis — A linear mixed effects model tested the interaction between group and condition on Q0 (derived intensity). Results: Condition: X2(6) = 6.59, p = 0.36 Group: X2(1) = 0.07, p = 0.79 Condition:Group: X2(6) = 7.38, p = 0.29
Statistical Analysis 2: Comparison: Exclusive Cigarette Smokers vs Dual Cigarette/ Nicotine Vaping Product Users; Test type: Other; p = 0.46, Mixed Models Analysis — A linear mixed effects model tested the interaction between group and condition on Alpha (demand elasticity). Results: Condition: X2(6) = 0.0001, p = 1.00 Group: X2(1) = 0.00, p = 0.99 Condition:Group: X2(6) = 5.65, p = 0.46

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Exclusive Cigarette Smokers | Dual Cigarette/ Nicotine Vaping Product Users
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT05177848/Prot_SAP_000.pdf